CLINICAL TRIAL: NCT05030311
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study of Remibrutinib (LOU064) to Investigate the Efficacy, Safety and Tolerability for 52 Weeks in Adult Chronic Spontaneous Urticaria (CSU) Patients Inadequately Controlled by H1-antihistamines
Brief Title: A Phase 3 Study of Efficacy and Safety of Remibrutinib in the Treatment of CSU in Adults Inadequately Controlled by H1 Antihistamines
Acronym: REMIX-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOU064A2301; 2022-001034-11 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-09-01 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: BTK inhibitor; Chronic spontaneous urticaria; Urticaria activity score; Hives severity score; Itch severity score; CSU
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LOU064 25mg b.i.d. (Experimental): Patients initially randomized to Remibrutinib during the Double-blind treatment period and continued Remibrutinib during the Open-label treatment period (Up to Week 52)
  Interventions: Drug: LOU064 25 mg (b.i.d); Drug: LOU064 25 mg (b.i.d) as a tablet.
- Placebo (Placebo Comparator): Patients initially randomized to Placebo (Up to Week 24)
  Interventions: Drug: Placebo; Drug: LOU064 25 mg (b.i.d) as a tablet.

INTERVENTIONS:
Drug: LOU064 25 mg (b.i.d) — LOU064 25 mg was administered by oral route twice a day (b.i.d) as a tablet.
  Other Names: remibrutinib
  Arms: LOU064 25mg b.i.d.
Drug: Placebo — Placebo
  Arms: Placebo
Drug: LOU064 25 mg (b.i.d) as a tablet. — LOU064 25 mg was administered by oral route twice a day (b.i.d) as a tablet in open label phase.
  Other Names: remibrutinib

SUMMARY:
The purpose of this study was to establish the efficacy, safety, and tolerability of remibrutinib (LOU064) in adult participants suffering from chronic spontaneous urticaria (CSU) inadequately controlled by H1-antihistamines in comparison to placebo.

DETAILED DESCRIPTION:
This was a global Phase III multi-centered, randomized,double-blind, parallel-group, placebo-controlled study investigating the safety, tolerability, and efficacy of remibrutinib (25 mg b.i.d.) in adult patients with CSU inadequately controlled by second generation H1-antihistamines (H1-AHs). The study consisted of four periods, the total study duration was up to 60 weeks: Screening period of up to 4 weeks, Double-blind placebo-controlled treatment period of 24 weeks, Open-label treatment period with remibrutinib period of 28 weeks, and treatment-free follow-up period of 4 weeks. The planned sample size was approximately 450 patients randomized in 2:1 ratio to remibrutinib or placebo arm (300 in the remibrutinib arm and 150 in placebo arm).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male and female adult participants ≥18 years of age.
* CSU duration for ≥ 6 months prior to screening (defined as the onset of CSU determined by the investigator based on all available supporting documentation).
* Diagnosis of CSU inadequately controlled by second generation H1 antihistamines at the time of randomization defined as:
* The presence of itch and hives for ≥6 consecutive weeks prior to screening despite the use of second generation H1-antihistamines during this time period
* UAS7 score (range 0-42) ≥16, ISS7 score (range 0-21) ≥ 6 and HSS7 score (range 0-21) ≥ 6 during the 7 days prior to randomization (Day 1)
* Documentation of hives within three months before randomization (either at screening and/or at randomization; or documented in the participants medical history).
* Willing and able to complete an Urticaria Patient Daily Diary (UPDD) for the duration of the study and adhere to the study protocol.
* Participants must not have had more than one missing UPDD entry (either morning or evening) in the 7 days prior to randomization (Day 1).

Exclusion Criteria:

* Participants having a clearly defined predominant or sole trigger of their chronic urticaria (chronic inducible urticaria) including urticaria factitia (symptomatic dermographism), cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic-, or contact-urticaria
* Other diseases with symptoms of urticaria or angioedema, including but not limited to urticaria vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary urticaria, or drug-induced urticaria
* Any other skin disease associated with chronic itching that might influence in the investigator's opinion the study evaluations and results, e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or psoriasis
* Evidence of clinically significant cardiovascular (such as but not limited to myocardial infarction, unstable ischemic heart disease, New York heart association (NYHA) Class III/IV left ventricular failure, arrhythmia and uncontrolled hypertension within 12 months prior to Visit 1), neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant
* Significant bleeding risk or coagulation disorders
* History of gastrointestinal bleeding, e.g. in association with use of nonsteroidal anti-inflammatory drugs (NSAID), that was clinically relevant (e.g. requiring hospitalization or blood transfusion)
* Requirement for anti-platelet medication, except for acetylsalicylic acid up to 100 mg/d or clopidogrel. The use of dual anti-platelet therapy (e.g. acetylsalicylic acid + clopidogrel) is prohibited.
* Requirement for anticoagulant medication (for example, warfarin or Novel Oral Anti-Coagulants (NOAC))
* History or current hepatic disease including but not limited to acute or chronic hepatitis, cirrhosis or hepatic failure or Aspartate Aminotransferase (AST)/ Alanine Aminotransferase (ALT) levels of more than 1.5 x upper limit of normal (ULN) or International Normalized Ratio (INR) of more than 1.5 at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (102):
- United States (26):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, North Little Rock, Arkansas
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Lancaster, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Redwood City, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Aventura, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Albany, Georgia
  - Novartis Investigative Site, Woodstock, Georgia
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Chevy Chase, Maryland
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Athens, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sandy City, Utah
  - Novartis Investigative Site, Bellingham, Washington
- Argentina (8):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Nueve De Julio
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Bahía Blanca
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Santa Fe
- Australia (3):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Bulgaria (2):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Colombia (4):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Czechia (4):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
- France (6):
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
- Hungary (3):
  - Novartis Investigative Site, Debrecen, Hajdú-Bihar
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- India (8):
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Belgavi
  - Novartis Investigative Site, Chandigarh
- Italy (4):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Torino, TO
- Japan (7):
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Villahermosa, Tabasco
- Puerto Rico (2):
  - Novartis Investigative Site, Carolina
  - Novartis Investigative Site, San Juan
- Novartis Investigative Site, Izhevsk, Russia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (6):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (6):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kayseri
  - Novartis Investigative Site, Sakarya
  - Novartis Investigative Site, Samsun
  - Novartis Investigative Site, Talas Kayseri

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Metz M, Gimenez-Arnau A, Hide M, Lebwohl M, Mosnaim G, Saini S, Sussman G, Szalewski R, Haemmerle S, Lheritier K, Martzloff ED, Seko N, Wang P, Zharkov A, Maurer M; REMIX-1 and REMIX-2 Investigators; REMIX-1 Investigators; REMIX-2 Investigators. Remibrutinib in Chronic Spontaneous Urticaria. N Engl J Med. 2025 Mar 6;392(10):984-994. doi: 10.1056/NEJMoa2408792. PMID 40043237
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2429

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted globally across 18 countries. Participants underwent a screening period of up to 4 weeks.
Period: Overall Study
Arm/Group | LOU064 25mg b.i.d. | Placebo
Started (All randomized patients, regardless of whether or not they received a dose of study drug.) | 313 | 157
Safety Set (All patients who received at least one dose of study treatment, whether or not randomized.) | 309 | 153
Full Analysis Set (FAS) (All patients to whom study treatment was assigned by randomization. Mis-randomized patients were excluded from FAS.) | 309 | 153
Completed | 251 | 124
Not Completed | 62 | 33
Not completed — Technical problems | 0 | 1
Not completed — Withdrawal by Subject | 31 | 17
Not completed — Adverse Event | 13 | 5
Not completed — Unsatisfactory therapeutic effect | 4 | 3
Not completed — Physician Decision | 5 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Protocol Violation | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LOU064 25mg b.i.d. | Placebo | Total
Number analyzed (Participants) | 313 | 157 | 470
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (14.27) | 45.9 (13.44) | 45 (13.99)
Age, Customized [Count of Participants; unit: Participants]
  >= 18 - < 65 years | 282 | 143 | 425
  >= 65 - < 85 years | 31 | 14 | 45
  >= 85 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 109 | 321
  Male | 101 | 48 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 44 | 120
  Not Hispanic or Latino | 237 | 113 | 350
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 14 | 26
  Asian | 94 | 46 | 140
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 3 | 15
  White | 188 | 89 | 277
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Urticaria Score (UAS7) at Week 12 (Scenario 1 With UAS7 as Primary Efficacy Endpoint)
Description: The Weekly Urticaria Activity Score (UAS7) is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42 (highest urticaria severity), and a minimum possible score of 0.
  This endpoint is a secondary endpoint for testing strategy Scenario 2 with Weekly Itch Severity Score (ISS7) and Weekly Hives Severity Score (HSS7) as co-primary efficacy endpoints).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
Scores on a scale | -20.02 (0.716) | -13.79 (0.980)
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -6.22, 95% CI 2-sided [-8.45 to -4.00], Standard Error of Mean 1.136 — MMRM adjusting for treatment arm, geographical region, prior exposure to anti-IgE biologics, visit week, baseline score and both interaction of treatment by visit week and interaction of baseline score by visit week

2. Primary Outcome: Change From Baseline in Weekly Itch Severity Score (ISS7) at Week 12 (Scenario 2 With ISS7 and HSS7 as Co-primary Efficacy Endpoints)
Description: The severity of the itch was recorded by the participant twice daily in their electronic Diary, on a scale of 0 (none) to 3 (severe). A weekly score (ISS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest itch severity).
  This endpoint is a secondary endpoint for testing strategy Scenario 1 with Weekly Urticaria Activity Score (UAS7) as the primary efficacy endpoint).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
Scores on a scale | -9.52 (0.343) | -6.89 (0.470)
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; ISS7 at Week 12 (Scenario 2 with ISS7 and HSS7 as co-primary efficacy endpoints); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-3.70 to -1.56], Standard Error of Mean 0.544 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline in Weekly Hives Severity Score (HSS7) at Week 12 (Scenario 2 With ISS7 and HSS7 as Co-primary Efficacy Endpoints)
Description: The hives (wheals) severity score, defined by number of hives, was recorded by the participant twice daily in their electronic Diary, on a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly score (HSS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest hives activity).
  This endpoint is a secondary endpoint for testing strategy Scenario 1 with Weekly Urticaria Activity Score (UAS7) as the primary efficacy endpoint.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
Scores on a scale | -10.47 (0.401) | -6.86 (0.548)
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; HSS7 at Week 12 (Scenario 2 with ISS7 and HSS7 as co-primary efficacy endpoints); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.61, 95% CI 2-sided [-4.85 to -2.36], Standard Error of Mean 0.635 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Patients Who Achieved Disease Activity Control (UAS7 ≤6)
Description: The percentage of patients achieving disease activity control (UAS7 =< 6) at Week 12 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
Participants | 154 | 38
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; Disease activity control (UAS7 =< 6) at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic; Logistic regression adjusting for treatment arm, geographical region, prior exposure to anti-IgE biologics, and baseline UAS7 score; Odds Ratio (OR) = 3.11, 95% CI 2-sided [2.00 to 4.84]

5. Secondary Outcome: Number of Patients Who Achieved Complete Absence of Hives and Itch (UAS7 = 0)
Description: The number of patients achieving complete absence of hives and itch (UAS7 = 0) at Week 12 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
Participants | 96 | 16
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; Complete absence of hives and itch (UAS7 = 0) at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 3.83, 95% CI 2-sided [2.16 to 6.82]

6. Secondary Outcome: Number of Patients With Early Onset of Disease Control (UAS7 ≤ 6 at Week 2)
Description: The percentage of patients achieving disease activity control (UAS7 =< 6) at Week 2 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 2
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
Participants | 104 | 5
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 15.67, 95% CI 2-sided [6.18 to 39.77] — Statistical model used logistic regression adjusting for treatment arm, geographical region, prior exposure to anti-IgE biologics, and baseline UAS7 score

7. Secondary Outcome: Cumulative Number of Weeks With Disease Activity Control (UAS7 <= 6) up to Week 12
Description: Maintaining disease activity control was assessed as cumulative number of weeks with an UAS7 =< 6 response between baseline and Week 12. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: up to Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: weeks
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
weeks | 5.17 (0.414) | 1.92 (0.241)
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; Test type: Superiority; p < 0.001, Negative binomial regression model; Negative binomial regression model with log link, using treatment arm, geographical region, and prior exposure to anti-IgE biologics as covariates; Rate ratio = 2.69, 95% CI 2-sided [2.01 to 3.61]

8. Secondary Outcome: Number of Patients Who Achieved DLQI = 0 - 1
Description: The Dermatology Life Quality Index (DLQI) is a 10-item (grouped in 6 domains) dermatology-specific quality of life (QoL) measure. Participants are rating their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse disease-related QoL). Domain scores are calculated for: Symptoms and Feelings (0-6), Daily Activities (0-6), Leisure (0-6), Work and School (0-3), Personal Relationships (0-6), Treatment (0-3). The overall DLQI score range was split into score bands and validated in terms of their meaning/relevance to patients overall. DLQI = 0-1 means no effect on patient's life.
Time Frame: Week 12
Population: Full Analysis Set (FAS) - for patients with a valid measurement without a protocol deviation with impact.
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 308 | 153
Participants | 120 | 34
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.53 to 3.90] — Statistical model used logistic regression adjusting for treatment arm, geographical region, prior exposure to anti-IgE biologics and baseline DLQI score

9. Secondary Outcome: Cumulative Number of Weeks Without Angioedema (AAS7 = 0)
Description: Angioedema occurrence was recorded once daily in the evening in the electronic Diary by the participant. Reporting the occurrence of angioedema was used as opening question for the assessment of the Angioedema Activity Score (AAS). The AAS consists of 5 questions with 4 answer options (scored 0-3) for each item, with a minimum score of 0 and a maximum score of 15 per day. The AAS score over 7 days (AAS7) ranges from 0 (no angioedema episodes) to 105 (highest angioedema severity).
Time Frame: Up to Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Weeks
Arm/Group | LOU064 25mg b.i.d. | Placebo
Number analyzed (Participants) | 309 | 153
Weeks | 8.43 (0.274) | 6.72 (0.330)
Statistical Analysis 1: Comparison: LOU064 25mg b.i.d. vs Placebo; Angioedema occurrence-free weeks (AAS7 = 0 response) up to Week 12; Test type: Superiority; p < 0.001, Regression, Linear; Rate ratio = 1.25, 95% CI 2-sided [1.12 to 1.41] — Statistical model used a negative binomial regression with log link included treatment arm as fixed effect, geographical region, prior exposure to anti-IgE biologics, baseline AAS7 = 0 response as covariates

10. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
Time Frame: On-treatment adverse events are reported from first dose of study medication up to 28 days after last dose of study medication, for a timeframe up to approximately 56 weeks
Population: Safety Set (SAF)
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind Treatment Period: LOU064 25 mg b.i.d.: Patients initially randomized to Remibrutinib (Up to Week 24)
- Double-blind Treatment Period: Placebo: Patients initially randomized to Placebo (Up to Week 24)
- Entire Study Period: LOU064 25mg b.i.d.: Patients initially randomized to Remibrutinib during the Double-blind treatment period and continued Remibrutinib during the Open-label treatment period (Up to Week 52)
- Open-label Period: Transitioned to LOU064 25 mg b.i.d.: Patients initially randomized to placebo during the Double-blind treatment period and switched to Remibrutinib during the Open-label treatment period (Weeks 25-52)
Arm/Group | Double-blind Treatment Period: LOU064 25 mg b.i.d. | Double-blind Treatment Period: Placebo | Entire Study Period: LOU064 25mg b.i.d. | Open-label Period: Transitioned to LOU064 25 mg b.i.d.
Number analyzed (Participants) | 309 | 153 | 309 | 133
Participants
  Patients with at least one AE | 188 | 86 | 218 | 62
  Patients with serious or other significant events - Death | 0 | 0 | 0 | 0
  Patients with serious or other significant events - SAEs | 10 | 1 | 13 | 1
  Discontinued study treatment due to any AEs | 11 | 3 | 15 | 2
  Patients with serious or other significant events - Discontinued study treatment due to any SAEs | 2 | 0 | 3 | 1
  Patients with serious or other significant events - Treatment interruption due to AEs | 17 | 9 | 18 | 3
  Patients with serious or other significant events - Treatment interruption due to SAEs | 5 | 1 | 5 | 0

ADVERSE EVENTS:
Time Frame: On-treatment adverse events are reported from first dose of study medication up to 28 days after last dose of study medication, for a timeframe up to approximately 56 weeks
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Groups:
- Transitioned to LOU064 25mg b.i.d.: Patients initially randomized to placebo during the Double-blind treatment period and switched to Remibrutinib during the Open-label treatment period (Weeks 25-52)
Arm/Group | LOU064 25mg b.i.d. | Placebo | Transitioned to LOU064 25mg b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/309 | 0/153 | 0/133
Serious Adverse Events (participants affected / at risk) | 13/309 | 1/153 | 1/133
Other Adverse Events (participants affected / at risk) | 139/309 | 53/153 | 26/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 25mg b.i.d. (N=309) | Placebo (N=153) | Transitioned to LOU064 25mg b.i.d. (N=133)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 25mg b.i.d. (N=309) | Placebo (N=153) | Transitioned to LOU064 25mg b.i.d. (N=133)
Diarrhoea (Gastrointestinal disorders) | 11 | 7 | 2
Nausea (Gastrointestinal disorders) | 11 | 3 | 0
Pyrexia (General disorders) | 10 | 3 | 1
COVID-19 (Infections and infestations) | 31 | 14 | 6
Influenza (Infections and infestations) | 10 | 2 | 4
Nasopharyngitis (Infections and infestations) | 22 | 5 | 6
Upper respiratory tract infection (Infections and infestations) | 12 | 2 | 3
Urinary tract infection (Infections and infestations) | 17 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 2
Headache (Nervous system disorders) | 25 | 11 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 11 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 11 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT05030311/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT05030311/SAP_001.pdf